CLINICAL TRIAL: NCT04505202
Title: Effect of Chlorhexidine-Induced Oral Care on Ventilator-Related Some Respiratory System Complications in Patients With Mechanical Ventilation
Brief Title: Effect of Chlorhexidine-Induced Oral Care on Ventilator-Related Some Respiratory System Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Duygu Kes, Principal Investigator, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2091
Record Dates: First submitted 2020-07-30; First posted 2020-08-10 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Ventilator Associated Pneumonia; Tracheobronchitis
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — chlorhexidine gluconate; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 0.12% chlorhexidine gluconate
  Interventions: Drug: 0.12% chlorhexidine gluconate
- Placebo group (Placebo Comparator): sodium bicarbonate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.12% chlorhexidine gluconate — The patients included in the experimental group (0.12% chlorhexidine gluconate) will receive 3 times daily oral care
  Arms: Experimental group
Drug: Placebo — The patients included in the placebo group ( sodium bicarbonate) will receive 3 times daily oral care
  Other Names: sodium bicarbonate
  Arms: Placebo group

SUMMARY:
Ventilator-associated pneumonia and ventilator-associated treakeabronchitis in respiratory tract infections associated with ventilator are common infections in intensive care unit and cause significant morbidity, mortality and health expenditures in nosocomial infections. Adequate and effective oral care by nurses in intensive care patients, possible complications, intensive care unit stay in the intensive care unit and is very important in terms of mortality.

DETAILED DESCRIPTION:
The aim of this study will (1) evaluate the effect of 0.12% chlorhexidine gluconate on ventilator-associated pneumonia, ventilator-associated treakeabronchitis, (2) determine the effect of preventing microorganism colonization, and (3) assess the mortality rate for each patient and the cost-effectiveness in the health expenditures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission in critical care with in 24 hours
* Having an endotracheal tube

Exclusion Criteria:

* History of chlorhexidine allergy
* Duration of mechanichal ventilation less than 48 h
* Confirmed diagnosis of pneumonitis before admission in the ICU
* Transfer from another ICU
* Receiving chemotherapy or radiotherapy
* Patients with immunodeficiency
* Patients with tracheostomies
* Required specific oral hygiene procedures
* Facio-maxillary or dental trauma/surgery
* Being pregnant

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Pathogen colonization change | change from baseline pathogen colonization at Day 3
  We will examine microbiological analyses ( mini-BAL, oropharyngeal and tracheal secretions)
Oral assessment guide score change | at the time of admission into the study (day 0), at study day 2 and at day 3
  The score ranges from 8 to 24 and higher scores indicating worse oral health
Clinical pulmonary infection score change | at the time of admission into the study (day 0), at study day 2 and at day 3
  The score ranges from 0 to 12 (ventilator-associated pneumonia ≥ 6 )
rate of tracheobronchitis change | change from baseline the rate of tracheobronchitis at Day 3
  Questionary (use the rate of tracheobronchitis categories)

SECONDARY OUTCOMES:
cost effectiveness | Day 30
  We used the decision tree modelling for estimating the cost-effectiveness of antiseptic solutions.
Mortality | Day 7 and Day 28
  rate of mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Karabük University Training and Research Hospital, Karabük, Karabük Province, Turkey (Türkiye)